CLINICAL TRIAL: NCT04587817
Title: An Observational, Single-center Study of Radiotherapy Combined With Immunotherapy for Massive Tumors
Brief Title: Combination of Hyperfractionated Radiotherapy With Immunotherapy in Massive Tumors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xian-shu Gao, Professor, Peking University First Hospital
Other Study IDs: 20200915
Record Dates: First submitted 2020-09-15; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Immunotherapy; SBRT; Bulky Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Camrelizumab+Hypofractionated radiation therapy: Camrelizumab: 200mg every 2 weeks until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment.
  Hypofractionated Radiotherapy(SABR): tumor center dose of 24-32Gy/8Gy/3-4f and surrounding important organs at risk ≤3.0Gy will be performed when one week following completion of the first immunotherapy. And the routine radiotherapy will be started with reaching a radical cure dose for the tumor margin. Generally, the radiotherapy will end before the fourth immunotherapy.
  Interventions: Combination Product: camrelizumab+hyperfractionated radiotherapy

INTERVENTIONS:
Combination Product: camrelizumab+hyperfractionated radiotherapy — Immunotherapy combined with hyperfractionated radiotherapy

SUMMARY:
This trial will explore effectiveness and safety using the combination therapy of camrelizumab and hyperfractionated radiotherapy in patients with massive tumor including non-small cell lung cancer, soft tissue sarcoma or urothelial carcinoma. Hypofractionation which represented by stereotactic body radiation therapy (SBRT) is a technique that delivers higher daily doses of radiation over a shorter period of time. This trial will also observe the index which can influencing the curative effect of hyperfractionated radiotherapy combined with immunotherapy.

DETAILED DESCRIPTION:
This trial is a prospective, observational, single-center, single-arm clinical research. This trial will explore effectiveness and safety using the combination therapy of camrelizumab and hyperfractionated radiotherapy in patients with massive tumor including non-small cell lung cancer, soft tissue sarcoma or urothelial carcinoma. All enrolled patients will receive the following treatments: camrelizumab 200mg every 2 weeks until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment. One week following completion of the first immunotherapy, hypofractionated radiotherapy(SABR) with tumor center dose of 24-32Gy/8Gy/3-4f and surrounding important organs at risk ≤3.0Gy will be performed. And the routine radiotherapy will be started with reaching a radical cure dose for the tumor margin. Generally, the radiotherapy will end before the fourth immunotherapy.

During treatment participants will be assessed for curative effects and the occurrence of adverse events. Following treatment, participants will be assessed at a clinic visit every 3 months to collect survival information and follow-up treatment information. The planned sample size is 60 study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female；
2. ECOG score will be 0 - 2；
3. The life expectancy will be longer than 12 weeks；
4. Patients with non-small cell lung cancer, soft tissue sarcoma or urothelial carcinoma were confirmed by histopathology；
5. Contain at least 1 measurable lesion with the largest long diameter ≥ 5cm;
6. The main organ functions are normal, and the results of laboratory test must be met the following criteria: Absolute neutrophil count（ANC）: more than 1.5 × 109/L; Platelets（PLT）: more than 75× 109/L; Total Bilirubin（TBil）：less than the upper normal limit (ULN); ALT and AST：less than 2.5 folds of the upper normal limit (ULN)，if there is liver metastasis, ALT and AST must be less than 5 folds of the upper normal limit (ULN) ; Urea Nitrogen (BUN): less than 2.5×ULN；Endogenous creatinine clearance ≥45 ml/min (Cockcroft-Gault formula);
7. Female subjects of childbearing age must undergo a serum pregnancy test within 3 days before starting the study drug, and the result is negative.Female and male subjects should take effective contraceptive measures from the beginning of treatment to within 3 months after the end of treatment;
8. Agreeing to participate in this study and signing a written informed consent.

Exclusion Criteria:

1. Central nervous system metastasis (including brain metastasis, meningeal metastasis, etc.);
2. Other immunosuppressive drugs used within 14 days before before study drug administration, excluding nasal sprays and inhaled corticosteroids or physiological doses of systemic steroids (ie not more than 10 mg/day of prednisolone or Other corticosteroids of equivalent pharmacological physiological dose);
3. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents: systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥ 90 mmHg;
4. Clinically significant cardiovascular diseases：Myocardial ischemia or myocardial infarction above grade II, ventricular arrhythmia which poorly controlled，QTc>450ms（male）/QTc>470ms (female)；Congestive heart failure (New York heart association (NYHA) class is Ⅲ～Ⅳ)；or cardiac color Doppler ultrasound examination revealed that the left ventricular ejection fraction (LVEF) <50%;
5. Accompanied by uncontrolled pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
6. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism;
7. Asthma that requires intermittent use of bronchodilators or other medical intervention should be excluded（Asthma has been completely relieved in childhood, and those without any intervention after adulthood can be included);
8. Coagulation abnormalities (INR>1.5、PT>ULN+4s、APTT >1.5 ULN）, with bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
9. Proteinuria ≥ (++) and 24 hours total urine protein > 1.0 g;
10. Received major surgery or suffered severe traumatic injury, fracture or ulcer within 4 weeks before enrollment;
11. Severe infections (such as intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks before the first administration, or unexplained fever> 38.5°C during the screening period/before the first administration;
12. Clinically significant hemoptysis or more than half a teaspoon (2.5ml) of hemoptysis per day occurred within 2 months before enrollment; or Clinically significant bleeding symptoms or tendency, such as gastrointestinal bleeding, hemorrhagic Gastric ulcer, fecal occult blood≥++ at baseline, or vasculitis, etc.;
13. Arterial/venous thrombosis events occurred in the 12 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
14. History of immunodeficiency or human immunodeficiency virus (HIV) infection, HBV DNA>500 IU/ml, HCV RNA>1000copies/ml, HBsAg+ and anti-HCV+；
15. Patients with a clear history of allergies may be potentially allergic or intolerant to camrelizumab and apatinib;
16. Patients who have a history of psychotropic drug abuse and cannot be quit or have mental disorders;
17. Other condition, illness, psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or stereotactic radiotherapy administration, or may interfere with the interpretation of study results and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous sampling was performed in the Department of Radiotherapy, Peking University First Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2022-09-19 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  The date of first treatment until the date of progression using the RECIST 1.1 criteria, or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Subject safety | 2 years
  Number of Adverse Events using NCI CTCAE 5.0
Overall Survival(OS) | 2 years
  Overall survival, defined from the date of first treatment to the date of death due to any cause.
Objective response rate(ORR) | 2 years
  Objective response rate, which is defined as the proportion of subjects who achieve a best response of complete response (CR) or partial response (PR) using the RECIST 1.1 criteria.
Disease control rate(DCR) | 2 years
  Disease control rate, which is defined as the proportion of subjects who achieve a response of complete response，partial response and stable disease (PR+CR+SD) in the total number of evaluable subjects using the RECIST 1.1 criteria
Local Control Rate | 2 years
  Local Control Rate, which is defined as the proportion of subjects who achieve a response of remission and stable disease (PR+CR+SD) evaluated by RECIST 1.1 after radiotherapy
Distant metastasis-free survival(DMFS) | 2 years
  Distant metastasis-free survival(DMFS), defined from the date of first treatment to the date of the appearance of distant metastasis or death due to any cause.
Response rate of lesions that did not receive radiotherapy | 2 years
  Response rate of lesions that did not receive radiotherapy, which is defined as the percentage of the number of cases with tumors that have not received radiotherapy in remission and stable disease (PR+CR+SD) in the total number of evaluable cases using the RECIST 1.1 criteria.
Quality of Life: EORTC QLQ-C30 questionnaire | 2 years
  Quality of life, which will be evaluated using the EORTC（The European Organization for Reasearch and Treatment of Cancer) QLQ-C30（Quality of Life Questionnare-Core 30） questionnaire. The questionnaire contains 30 items. Items 29 and 30 are divided into seven levels, which are counted from 1 to 7 points, 1 is very poor, and 7 is very good. Other items are divided into 4 levels: no at all, a little bit, a lot, and very, and they are directly rated from 1 to 4 points

CONTACTS AND LOCATIONS:
Overall Officials: Xianshu Gao, MD,PhD, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No